CLINICAL TRIAL: NCT07275099
Title: Quality of Life, Psychological Impact and Care-related Challenges in Patients Affected by Von Hippel-Lindau Syndrome: a Single-centre Observational, Transversal, Study.
Brief Title: Quality of Life, Psychological Impact, and Care-related Challenges in Patients Affected by Von Hippel-Lindau Syndrome.
Acronym: QoL- VHL
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Larcher Alessandro, Medical Doctor, IRCCS Ospedale San Raffaele
Other Study IDs: QoL- VHL
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-10

CONDITIONS: VHL - Von Hippel-Lindau Syndrome
MeSH Terms: conditions — von Hippel-Lindau Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single - centre, cross - sectional observational study with additional procedure.: Adult subjects (≥ 18 years) with confirmed diagnosis of von Hippel - Lindau syndrome

SUMMARY:
This is a single-centre, cross-sectional observational study aiming to assess the psychological burden, quality of life, and perceived barriers to care in patients with von Hippel-Lindau syndrome (VHL). Data will be collected through an anonymous online questionnaire, specifically designed for the study and administered via Google Forms.

DETAILED DESCRIPTION:
This is a single-centre, cross-sectional observational study designed to assess the psychological burden and health-related quality of life in individuals with von Hippel-Lindau (VHL) syndrome, and to explore perceived barriers to healthcare access and the perceived adequacy of multidisciplinary care.

The hypothesis underlying this study is that individuals affected by VHL experience a substantial psychological burden and face variable access to appropriate care pathways, which may differ based on demographic or clinical factors.

The study will involve a single group of participants (n ≈ 200). No control group or randomization is foreseen. The study duration is estimated at 10 years, including data collection and analysis.

Each participant will be involved once, with a single data collection session (approx. 25-30 minutes) through the study-specific questionnaire "VHL: Accesso alle cure e vita quotidiana". The questionnaire, administered in Italian via the Google Forms platform, is not part of routine clinical practice and is administered exclusively for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Genetically confirmed diagnosis of von Hippel- Lindau syndrome

Exclusion Criteria:

* Inability to understand or complete the questionnaire, either independently or with assistance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects (≥18 years) with confirmed diagnosis of von Hippel - Lindau syndrome
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2035-12-01 (Estimated); Study Completion 2035-12-01 (Estimated)

PRIMARY OUTCOMES:
Completion of a self- administered questionnaire | Single time point (approximately 25-30minutes).
  The research activity consists in the anonymous collection of patient- reported data through an online questionnaire. No diagnostic, therapeutic, or experimental interventions are foreseen. The study fully complies with the definition of non-interventional observational research.